CLINICAL TRIAL: NCT06646939
Title: Comparison of Community Reintegration Interventions Relative to the Institution of a Simulated Environment in Inpatient Rehabilitation and Pilot Study of the Impact of Simulated Environment on Functional Outcomes
Brief Title: Comparison of Community Reintegration Interventions When Using a Simulated Environment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hunter College of The City University of New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-07025042
Record Dates: First submitted 2024-10-02; First posted 2024-10-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Simulated Environments for Community Reintegration
Keywords: Inpatient Rehabilitation Unit; Community Reintegration; Simulated Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Reintegration in Simulated Environment (Experimental)
  Interventions: Behavioral: PT and OT with a simulated environment

INTERVENTIONS:
Behavioral: PT and OT with a simulated environment — Upon admission to the inpatient rehabilitation unit, participants will undergo a physical and occupational therapy evaluation. The evaluations will include the outcome measures chosen to track for this study (10-meter walk test and Quality Indicators). If a patient meets inclusion/exclusion criteria, informed written consent will be obtained. Throughout the patient's stay, therapists will have the opportunity to perform community integration treatments using the simulated environment. This could include activities such as negotiating a curb, crossing a street, or shopping at a marketplace. The therapist will document the amount of time (units billed) spent performing these interventions. The research investigators will not act as a patient's therapist throughout their admission.

SUMMARY:
The investigators believe that rehabilitation specialists will use community reintegration treatments more if a simulated environment is available.

DETAILED DESCRIPTION:
Community reintegration training has always been a significant aspect of inpatient rehabilitation recovery. Community reintegration training involved therapists and patients going into the actual community to evaluate and practice their functional tasks such as negotiating curbs, crosswalks, or marketplaces. During the COVID-19 pandemic, this option was not available. The absence of this intervention made it challenging for therapists to evaluate a patient's safety to return home. Creating a simulated environment within the inpatient rehabilitation department became an alternative to taking patients to an outside environment. Saji, et al. (2015) demonstrated that utilization of a simulated environment enhanced functional improvements of post-acute stroke patients at 12 convalescent rehabilitation wards. New York Presbyterian Weill Cornell Medical Center (NYP- WCMC) has constructed a simulated environment for the purposes of enhancing community reintegration training. This project will test its use and efficacy.

The availability of this simulated environment may be more time-efficient and safer than community reintegration training outside of the department or hospital. Training in the simulated environment may improve the functional ability of individuals undergoing inpatient rehabilitation, in accordance with the degree of use of the simulated environment. Greater use of the simulated environment may predict greater functional improvements. This study will collect pilot data about functional outcomes and patient perspectives about their balance confidence, their ability to perform functional tasks, and the efficacy of the use of simulated environment for community reintegration. This pilot data will seed a future efficacy study with a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Medical records of patients admitted to the IRU from January 1, 2015 through December 31, 2019 will be queried for number of minutes billed for Community Integration.
* Medical records of patients admitted to the IRU from April 2
* Patients admitted to the Inpatient Rehabilitation Unit (IRU) of at least 18 years of age and older
* Patients who can read and provide informed consent in English.
* Patients who will be discharged to home after inpatient rehabilitation.
* Patients who are ambulatory with a minimal QI score of 3 on "Walk 10 feet".
* Patients who utilized the simulated environment during their inpatient stay.
* Patients who score 8 or greater on the BIMS on initial evaluation.

Exclusion Criteria:

* The investigators will exclude medical records of patients admitted to the IRU from January 1, 2020 through December 31, 2021 because of the COVID restrictions that were in place.
* Patients who are less than 18 years of age.
* Patients who are not ambulatory due to medical reasons.
* Patients who cannot read and provide informed consent in English.
* Patients who were discharged to acute care, skilled nursing facility or long-term care facility after their inpatient rehabilitation stay.
* Patients who did not use the simulated environment during their inpatient stay.
* Patients who score 7 or lower on the BIMS on initial evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Utilization of community reintegration, as measured by number of 15-minute units billed | Duration of IRU stay, an average of 11 days
  Current Procedural Terminology (CPT) code 9753, is a billing code where one unit of the code is used for each 15 minutes the provider spends with the patient teaching them return to work and the community.
  For this measure, the therapist will document the amount of time spent performing each study activity when utilizing the simulated environment, as measured by number of 15-minute units billed..
  This will be compared to units billed in 2015 - 2019 prior to the implementation of the simulated environment for this study.

SECONDARY OUTCOMES:
Quality Indicators | Duration of IRU stay, an average of 11 days
  Qualitative assessment by the therapist of 1 step onto and off a curb
Quality Indicators | Duration of IRU stay, an average of 11 days
  Qualitative assessment by the therapist of picking up an object
Quality Indicators | Duration of IRU stay, an average of 11 days
  Qualitative assessment by the therapist of walking 10 feet on uneven surface
Quality Indicators | Duration of IRU stay, an average of 11 days
  Qualitative assessment by the therapist of car transfer
Gait Speed | Duration of IRU stay, an average of 11 days
  Meters/second
Activities Specific Balance Confidence Scale | Duration of IRU stay, an average of 11 days
  The Activities-specific Balance Confidence (ABC) scale is scored by adding up the ratings for each item and dividing by 16, the total number of items.
  The scale uses a range of 0-100%, with 0 representing no confidence and 100 representing complete confidence.
  The resulting score indicates the participant's overall balance confidence. 80% or higher: The participant has a high level of physical functioning and is at low risk for falls 50-80%: The participant has a moderate level of physical functioning Less than 50%: The participant has a low level of physical functioning and is at a high risk of falling Less than 67%: The participant has a substantial risk of falling
Patient satisfaction | Date of Discharge (at approximately Day 11)
  Likert scale, with a low score of 1 and a high score of 5.
Patient satisfaction | 30 days post discharge
  Likert scale, with a low score of 1 and a high score of 5.
Length of Stay | Duration of IRU stay, an average of 11 days
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chowdhury, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork Presbyterian Hospital Baker Pavilion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohannon RW. Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants. Age Ageing. 1997 Jan;26(1):15-9. doi: 10.1093/ageing/26.1.15. PMID 9143432
- [Background] Saliba D, Buchanan J, Edelen MO, Streim J, Ouslander J, Berlowitz D, Chodosh J. MDS 3.0: brief interview for mental status. J Am Med Dir Assoc. 2012 Sep;13(7):611-7. doi: 10.1016/j.jamda.2012.06.004. Epub 2012 Jul 15. PMID 22796362
- [Background] Richardson J, Law M, Wishart L, Guyatt G. The use of a simulated environment (easy street) to retrain independent living skills in elderly persons: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2000 Oct;55(10):M578-84. doi: 10.1093/gerona/55.10.m578. PMID 11034230
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Peel NM, Kuys SS, Klein K. Gait speed as a measure in geriatric assessment in clinical settings: a systematic review. J Gerontol A Biol Sci Med Sci. 2013 Jan;68(1):39-46. doi: 10.1093/gerona/gls174. Epub 2012 Aug 24. PMID 22923430
- [Background] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Eyssen IC, Beelen A, Dedding C, Cardol M, Dekker J. The reproducibility of the Canadian Occupational Performance Measure. Clin Rehabil. 2005 Dec;19(8):888-94. doi: 10.1191/0269215505cr883oa. PMID 16323388
- See also: Braden H. Self-selected gait speed: A Critical clinical outcome. Lower Extremity Review Magazine. November, 2012. — https://lermagazine.com/article/self-selected-gait-speed-a-critical-clinical-outcome=